CLINICAL TRIAL: NCT03102164
Title: Evaluation of Skeletal Muscles During Acute Heart Failure
Brief Title: Skeletal Muscles in Acute Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Responsible Party: Principal Investigator, Kinga Węgrzynowska-Teodorczyk, PhD in physiotherapy, Wroclaw University of Health and Sport Sciences
Other Study IDs: UMO-2013/11/D/NZ7/00922
Record Dates: First submitted 2017-03-14; First posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Heart Decompensation
Keywords: heart failure; decompensation
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collection of blood samples for centrifugation, pipetting, frozing and the anaysis of ferritin, iron, albumin + protein + bilirubin, GGT, AST + ALT, hsCRP, NTproBNP, creatinine, complete blood count with smear creatine kinase + enzymes, CK-mass, venous blood gasometry
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cardiac rehabilitation: patients undergoing cardiologic rehabilitation according to the protocol used routinely at the Military Hospital in Wroclaw.The protocol of rehabilitation, adjusted to clinical status, individual needs and physical capability of the patient, includes gradually increasing level of physical exercise. Upon achieving relative stabilization of clinical status and excluding absolute contraindications to physical exercise, usually on the 2nd or 3rd day of hospitalization, the cardiologic rehabilitation is ordered by a physician in charge. The rehabilitation protocol comprises respiratory, assisted, active dynamic,and relaxation exercises, as well as short-term isometric exercises and general strength exercises of very low intensity, short duration and properly adjusted recovery phase;they are conducted in a lying, sitting, or standing position.
  Interventions: Procedure: cardiac rehabilitation
- Controls: patients treated using standard pharmacotherapy within Center for Heart Disease, Military Clinical Hospital in Wroclaw.

INTERVENTIONS:
Procedure: cardiac rehabilitation — The rehabilitation protocol comprises respiratory, assisted, active dynamic, and relaxation exercises, as well as short-term isometric exercises and general strength exercises of very low intensity, short duration and properly adjusted recovery phase; they are conducted in a lying, sitting, or standing position.
  Groups: cardiac rehabilitation

SUMMARY:
The study will include 30 consecutive patients with acute heart failure (AHF). In 20 patients the investigators will perform cardiologic rehabilitation. In the remaining 10 patients only standard pharmacotherapy will be administered. The cardiologic rehabilitation will follow the protocol used routinely in patients with AHF admitted to the Centre for Heart Disease,Military Hospital in Wroclaw. This protocol includes gradually increasing level of physical exercise (e.g.: respiratory exercises, assisted, active dynamic, and relaxation exercises, as well as short-term isometric exercises and general exercises of very low intensity, short duration and properly adjusted recovery phase).

The following tests will be conducted on the first and last day of hospitalization and 30 days following the discharge:

clinical evaluation (medical interview, routine physical examination, echocardiography, assessment of natriuretic peptides (NT-proBNP), basic laboratory tests with special emphasis on the inflammatory markers and renal and liver parameters); hemodynamic evaluation (i.e. non-invasive evaluation of cardiac output and systemic vascular resistance using of impedance cardiography); evaluation of biomarkers reflecting myocyte-damage (i.e. immunochemical measures of tissue-specific enzymatic isoforms, enabling to distinguish the markers of skeletal muscle damage vs. markers of myocardial injury - e.g. creatine kinase CK, its muscular isozyme CKMM, lactate dehydrogenase 5 LDH5, myoglobin, and carbonic anhydrase III, determined using test based on ELISA). On the first day of hospitalization, as well as on the first, third and last day of rehabilitation (the latter term corresponding to the last day of hospitalization as well) and also 30 days after the discharge, the following tests will be performed (both times: at rest and post-exercise): hemodynamic evaluation, the evaluation of skeletal muscle function (using surface electromyography (sEMG); maximum tonus of the muscles will be determined along with the level of muscular fatigability and its changes over time; the evaluation of muscle tissue perfusion (assessed on the basis of oxygenation level, with non-invasive, direct continuous recording of the perfusion in peripheral tissues by local tissue oximetry, measured by the near-infrared spectroscopy (NIRS). NIRS is based on the absorption of near-infrared waves by oxygenated and reduced haemoglobin. The levels of absorption reflect the degree of tissue oxygenation in a given area of microcirculation. Furthermore, a capillary gasometry (oxygen saturation and lactate concentration) will be determined). Moreover, two functional tests will be performed at the discharge and 30 days after the discharge: the 6-minute walk test and the 30-second "chair stand" test examining the strength endurance of the lower extremities (pertaining to repeated getting up from a chair over a period of 30 seconds).

DETAILED DESCRIPTION:
T1. Objective and hypotheses Acute heart failure (AHF) is associated with the disorders of peripheral perfusion, leading to injury of many vital organs. Consequently, each episode of AHF can have a form of multiple organ failure with potential injury and dysfunction of skeletal muscles; however, this latter issue has not been addressed in literature thus far. The aim of this project is to comprehensively evaluate the skeletal muscles (at a functional and tissue level) during acute heart failure. The following hypotheses will be verified:(1) Impaired perfusion of the muscles is reflected by their injury and significant functional abnormalities; (2) Early implemented motor rehabilitation improves perfusion and function of skeletal muscles; This study will demonstrate that skeletal muscles are involved as a component of AHF-related multiple organ failure.

Moreover, study will involve the analysis of the effect of physical exercise sessions on the hemodynamic parameters of patients with AHF (cardiac output, stroke volume, arterial blood pressure, and systemic vascular resistance); this question has not been addressed thus far.

Method The study will include 30 consecutive patients with AHF (resulting from the decompensation of chronic systolic HF). In the case of 20 patients the therapeutic process will include cardiologic rehabilitation, and only standard pharmacotherapy will be administered in another 10 patients. The cardiologic rehabilitation will follow the protocol for patients with AHF used routinely at the Center for Heart Disease, Military Clinical Hospital with Polyclinic in Wroclaw. The protocol includes gradually increasing level of physical exercise: respiratory, assisted, active dynamic, and relaxation exercises, as well as short-term isometric exercises and general strength exercises of very low intensity, short duration and properly adjusted recovery phase.

The following tests will be conducted on the first and last day of hospitalization and 30 days following the discharge:

Clinical evaluation - history taking, routine physical examination, echocardiography, determination of natriuretic peptides (NT-proBNP), basic laboratory tests with special emphasis on the inflammatory markers and renal and liver parameters.

Hemodynamic evaluation - non-invasive determination of cardiac output and systemic vascular resistance by means of impedance cardiography.

Evaluation of myocyte injury markers - immunochemical measurements of tissue-specific enzymatic isoforms will be taken in order to distinguish between the markers of skeletal muscle and myocardial injury. The biomarkers of muscular injury (e.g. creatine kinase CK, its muscular isozyme CKMM, lactate dehydrogenase 5 LDH5, myoglobin, and carbonic anhydrase III) will be determined in serum by means of ELISA.

Moreover, the following tests will be conducted at rest and post-exercise on the first day of hospitalization, as well as on the first, third and last day of rehabilitation (the latter term corresponding to the last day of hospitalization as well) and 30 days after the discharge:

Evaluation of skeletal muscle function will be conducted by means of surface electromyography (sEMG). Maximum tonus of the muscles will be determined along with the level of muscular fatigability and its changes over time. Moreover, two functional tests will be conducted at discharge from the hospital and 30 days thereafter: the 6-minute walk test and the 30-second "chair stand" test examining the strength endurance of the lower body (pertaining to repeated getting up from a chair over a period of 30 seconds).

Evaluation of muscle tissue perfusion (examined indirectly on the basis of oxygenation level) will be conducted with non-invasively by direct continuous recording of perfusion in peripheral tissues by local tissue oximetry, the so-called near-infrared spectroscopy (NIRS). NIRS is based on the absorption of near-infrared waves by oxygenated and reduced hemoglobin. The levels of absorption reflect the degree of tissue oxygenation in a given area of microcirculation. Furthermore, a capillary gasometry (oxygen saturation and lactate concentration) will be determined

ELIGIBILITY:
Inclusion Criteria:

* patients with acute heart failure (AHF - defined according to the ESC criteria-

Exclusion Criteria:

* lack of written informed consent
* acute coronary syndrome
* bacterial infection confirmed on the basis of clinical and laboratory criteria
* preexisting chronic respiratory failure
* necessity of mechanical ventilation
* significant arrhythmia and conductivity disorders
* anemia (hemoglobin < 9g%)
* active neoplastic process
* liver injury (AST, ALT > 3 x reference level)
* chronic kidney failure with creatinine clearance < 30 ml/min.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include 30 patients with acute heart failure (AHF - defined according to the ESC criteria- hospitalized at the Center for Heart Disease, Military Clinical Hospital with Polyclinic in Wroclaw and diagnosed with chronic systolic heart failure at least 6 months prior to the admission.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-04-21 (Actual); Primary Completion 2017-12-21 (Estimated); Study Completion 2018-07-07 (Estimated)

PRIMARY OUTCOMES:
reduction of muscle fatigue | 1,5 months
  We expect that patients from the intervention group will demonstrate reduced muscle fatigability as compared to the controls. Frequency (Hz) and amplitude (mV) of potentials assessed using EMG will serve as a measure of muscle fatigue.
improvement of respiratory muscle strength | 1,5 months
  We expect that patients from the intervention group will demonstrate improved respiratory muscle strength as compared to the controls. Maximal inspiratory and expiratory pressures [both in cm H2O] will serve as measures of respiratory muscle strength.
improvement of functional fitness | 1,5 months
  We expect that patients from the intervention group will demonstrate improved functional fitness as compared to the controls. Results of the six motor tasks in the "Senior Fitness Test" (time (sec.) in Up-and-go; number of repetitions in Chair stand and Arm curl, distance (cm) in Sit-and-reach and Back scratch and distance (m) in six-minute walk test) will serve as a measures of functional fitness.

CONTACTS AND LOCATIONS:
Overall Officials: Kinga Węgrzynowska-Teodorczyk, phd, Principal Investigator — University School of Physical Education
Locations (1):
- University School of Physical Education in Wroclaw, Wroclaw, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No